CLINICAL TRIAL: NCT05419570
Title: Ability of Short Time Low PEEP Challenge and Mini Fluid Challenge to Predict Fluid Responsiveness During Pancreaticoduodenectomy
Brief Title: Short Time Low PEEP Challenge and Mini Fluid Challenge
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, Medical Doctor, Istanbul Saglik Bilimleri University
Other Study IDs: 2021.01.31
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Intraoperative Care; Fluid Responsiveness
Keywords: Intraoperative monitoring; fluid therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing Pancreaticoduodenectomy
  Interventions: Other: Fluid Loading

INTERVENTIONS:
Other: Fluid Loading — Hemodynamic and ventilatory parameters will be recorded at five time points (T1 - T5). After baseline meausrements (T1), additional 5 cmH2O PEEP will be applied to patients for 30 seconds (short time low peep challenge, SLPC). Prior to PEEP lowering T2 measurement will be performed. T3 measurement will be performed one minute after PEEP is decreased to its initial value and will be recorded as the second baseline. Thereafter, 100 ml isotonic saline will be infused over one minute (MFC). T4 measurement will be performed one minute after MFC is completed,. Lastly, T5 measurement will be performed three minutes after additional 400 ml of isotonic saline is infused within 10 minutes to complete 500 ml of fluid loading.

SUMMARY:
Optimizing fluid therapy is one of the main concerns for anesthesiologists during the intraoperative period. It becomes even more important in high-risk long lasting surgeries as pancreaticoduodenectomy. Therefore evaluating fluid responsiveness prior to fluid loading is highly recommended. To the best of our knowledge there is no study comparing the abilities short time low PEEP challenge and mini fluid challenge in predicting fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy

Exclusion Criteria:

* Body mass index (BMI) > 35 kg / m2
* any ventricular dysfunction
* Crs < 35 ml / cmH2O
* valvular heart disease
* ASA score > 3
* cardiac arrhythmia
* history of lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Difference between the abilities of two methods to predict fluid responsiveness defined as an increase in stroke volume index >15% after fluid loading | one day
  Difference between the area under reciever operating characterisitcs curve of two methods

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Başakşehir Çam adn Sakura City Hospital, Istanbul
  - Başakşehir Çam and Sakura City Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdullah T, Gokduman HC, Bahar Ozbey N, Sarban O, Ali A, Gumus Ozcan F. Comparison of the ability of short time low PEEP challenge and mini fluid challenge to predict fluid responsiveness in patients undergoing open pancreaticoduodenectomy: an observational cohort study. Eur Rev Med Pharmacol Sci. 2024 Jun;28(12):3860-3870. doi: 10.26355/eurrev_202406_36463. PMID 38946384